CLINICAL TRIAL: NCT00346489
Title: Intermediate Term Outcomes of Intraoperative 5-Fluorouracil Versus Mitomycin c in Trabeculectomy Surgery.
Brief Title: Outcomes of Intraoperative 5-Fluorouracil Versus Mitomycin C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0409-60
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Glaucoma
Keywords: Trabeculectomy; 5-fluorouracil; Mitomycin C
MeSH Terms: conditions — Glaucoma | interventions — Fluorouracil; Mitomycin

INTERVENTIONS:
Drug: 5-fluorouracil
Drug: Mitomycin C

SUMMARY:
A clinical trial to establish the long term response of using intraoperative 5-fluorouracil (5-FU) versus mitomycin C (MMC) in trabeculectomy glaucoma surgery. Antiproliferative agents such as 5-fluorouracil and Mitomycin C have been used extensively in trabeculectomy surgery to improve the success of the surgery and prevent further visual loss and blindness in glaucoma patients.

DETAILED DESCRIPTION:
Glaucoma is a life-long progressive disease, and patients are living longer. Therefore, a long term full evaluation of the efficacy of intraoperative 5-FU and MMC needs to be performed to assess the true efficacy of MMC compared to 5-FU. We, therefore propose, a long-term prospective study of patients previously enrolled in the prospective study involving the evaluation of single intraoperative application of mitomycin C versus 5-fluorouracil in low to moderate risk glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Only patients deemed successful as 36 months will be included. These patients will have participated in the randomized prospective study trial comparing intraoperative 5-FU and mitomycin C in primary trabeculectomy.

Exclusion Criteria:

* Only patients deemed successful as 36 months will be included. These patients will have participated in the randomized prospective study trial comparing intraoperative 5-FU and mitomycin C in primary trabeculectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Pressure Control

SECONDARY OUTCOMES:
Mitomycin Complications

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Cantor, MD, Principal Investigator — IUPUI/Clarian
Locations (2):
- United States (2):
  - University Hospital and Outpatient Center, Indianapolis, Indiana
  - IU Eye at Carmel, Indianapolis, Indiana

REFERENCES:
- [Background] Skuta GL, Beeson CC, Higginbotham EJ, Lichter PR, Musch DC, Bergstrom TJ, Klein TB, Falck FY Jr. Intraoperative mitomycin versus postoperative 5-fluorouracil in high-risk glaucoma filtering surgery. Ophthalmology. 1992 Mar;99(3):438-44. doi: 10.1016/s0161-6420(92)31951-7. PMID 1565457
- [Background] Kitazawa Y, Kawase K, Matsushita H, Minobe M. Trabeculectomy with mitomycin. A comparative study with fluorouracil. Arch Ophthalmol. 1991 Dec;109(12):1693-8. doi: 10.1001/archopht.1991.01080120077030. PMID 1841578
- [Background] Palmer SS. Mitomycin as adjunct chemotherapy with trabeculectomy. Ophthalmology. 1991 Mar;98(3):317-21. doi: 10.1016/s0161-6420(91)32293-0. PMID 2023752
- [Background] Dunn JP, Seamone CD, Ostler HB, Nickel BL, Beallo A. Development of scleral ulceration and calcification after pterygium excision and mitomycin therapy. Am J Ophthalmol. 1991 Sep 15;112(3):343-4. doi: 10.1016/s0002-9394(14)76738-8. No abstract available. PMID 1882947
- [Background] Fluorouracil Filtering Surgery Study one-year follow-up. The Fluorouracil Filtering Surgery Study Group. Am J Ophthalmol. 1989 Dec 15;108(6):625-35. doi: 10.1016/0002-9394(89)90853-2. PMID 2688428
- [Background] Liebmann JM, Ritch R, Marmor M, Nunez J, Wolner B. Initial 5-fluorouracil trabeculectomy in uncomplicated glaucoma. Ophthalmology. 1991 Jul;98(7):1036-41. doi: 10.1016/s0161-6420(91)32180-8. PMID 1891210
- [Background] Lee DA, Hersh P, Kersten D, Melamed S. Complications of subconjunctival 5-fluorouracil following glaucoma filtering surgery. Ophthalmic Surg. 1987 Mar;18(3):187-90. PMID 3587857
- [Background] Knapp A, Heuer DK, Stern GA, Driebe WT Jr. Serious corneal complications of glaucoma filtering surgery with postoperative 5-fluorouracil. Am J Ophthalmol. 1987 Feb 15;103(2):183-7. doi: 10.1016/s0002-9394(14)74224-2. PMID 3812620
- [Background] Khaw PT, Sherwood MB, MacKay SL, Rossi MJ, Schultz G. Five-minute treatments with fluorouracil, floxuridine, and mitomycin have long-term effects on human Tenon's capsule fibroblasts. Arch Ophthalmol. 1992 Aug;110(8):1150-4. doi: 10.1001/archopht.1992.01080200130040. PMID 1386726
- [Background] Khaw PT, Doyle JW, Sherwood MB, Grierson I, Schultz G, McGorray S. Prolonged localized tissue effects from 5-minute exposures to fluorouracil and mitomycin C. Arch Ophthalmol. 1993 Feb;111(2):263-7. doi: 10.1001/archopht.1993.01090020117035. PMID 8431167
- [Background] Khaw PT, Doyle JW, Sherwood MB, Smith MF, McGorray S. Effects of intraoperative 5-fluorouracil or mitomycin C on glaucoma filtration surgery in the rabbit. Ophthalmology. 1993 Mar;100(3):367-72. doi: 10.1016/s0161-6420(93)31640-4. PMID 8460007
- [Background] Lanigan L, Sturmer J, Baez KA, Hitchings RA, Khaw PT. Single intraoperative applications of 5-fluorouracil during filtration surgery: early results. Br J Ophthalmol. 1994 Jan;78(1):33-7. doi: 10.1136/bjo.78.1.33. PMID 8110695
- [Background] Dietze PJ, Feldman RM, Gross RL. Intraoperative application of 5-fluorouracil during trabeculectomy. Ophthalmic Surg. 1992 Oct;23(10):662-5. PMID 1436965
- [Background] Egbert PR, Williams AS, Singh K, Dadzie P, Egbert TB. A prospective trial of intraoperative fluorouracil during trabeculectomy in a black population. Am J Ophthalmol. 1993 Nov 15;116(5):612-6. doi: 10.1016/s0002-9394(14)73204-0. PMID 8238222
- [Background] Smith MF, Doyle JW, Nguyen QH, Sherwood MB. Results of intraoperative 4 fluorouracil or low dose MMC supplementation on primary trabeculectomy surgery. Invest Ophthalmol & Visual Science. 1996,37;#3:S25(Abstract #108).
- [Background] Singh K, Mehta K, Shaikh NM, Tsai JC, Moster MR, Budenz DL, Greenfield DS, Chen PP, Cohen JS, Baerveldt GS, Shaikh S. Trabeculectomy with intraoperative mitomycin C versus 5-fluorouracil. Prospective randomized clinical trial. Ophthalmology. 2000 Dec;107(12):2305-9. doi: 10.1016/s0161-6420(00)00391-2. PMID 11097613
- [Background] Spaeth GL, Mutlukan E. The use of antimetabolites with trabeculectomy: a critical appraisal. J Glaucoma. 2001 Jun;10(3):145-51. doi: 10.1097/00061198-200106000-00001. PMID 11442174
- [Background] WuDunn D, Cantor LB, Palanca-Capistrano AM, Hoop J, Alvi NP, Finley C, Lakhani V, Burnstein A, Knotts SL. A prospective randomized trial comparing intraoperative 5-fluorouracil vs mitomycin C in primary trabeculectomy. Am J Ophthalmol. 2002 Oct;134(4):521-8. doi: 10.1016/s0002-9394(02)01627-6. PMID 12383808